CLINICAL TRIAL: NCT01420354
Title: Can a Spot Urine Replace or Improve 24 Hour Urine Collections in Kidney Stone Patients
Status: Terminated | Type: Observational
Why Stopped: The study was combined with our Urine and Stool Study (NCT01637506).
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: H08-02934
Record Dates: First submitted 2010-10-18; First posted 2011-08-19 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Kidney Stones
Keywords: Metabolic stones; kidney stones; renal calculi; metabolic evaluation
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine collected over 24 hour period
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will sought to determine if limited urine collections can provide similar or more informative data than standard 24-hour urine collections used to evaluate kidney stone formers.

DETAILED DESCRIPTION:
BACKGROUND Urinary stone disease is a common problem, causing significant morbidity and sometimes mortality. Stone disease affects 5-10% of the population during their lifetime and of these patients between 30-50% will have at least one recurrent episode.

Urinary stones arise due to crystallization and aggregation of supersaturated ion complexes in the urine. Depending on the concentration of various urinary constituents and the physicochemical characteristics of a given individual's urine (such as pH, volume, calcium citrate concentration etc.), different crystals may precipitate. Therefore therapy is tailored to the individual, based on stone composition and the results of the 24-hour urine collection. The majority of the stones are calcium based (calcium oxalate, calcium phosphate) while the remaining are comprised of uric acid, struvite, cystine or other substances.

While some stones can pass spontaneously, the majority will require some form of treatment, and more than 50% will require surgical intervention. Until the 1980s, treatment of upper urinary tract stones often involved extensive open surgical procedures5. With the introduction of extracorporeal shock-wave lithotripsy (ESWL) and refinements in endourological procedures like percutaneous nephrolithotomy (PCNL), ureteroscopy (URS) techniques, it has now become possible to treat stones in almost all cases without open surgery. Stone management can be divided into three treatment phases. The first phase involves treatment of acute pain and the drainage of an obstructed and possibly infected kidney. The second phase aims to either remove or disintegrate the stone. The third phase is directed towards the prophylaxis of stone recurrence .

The third phase involves the metabolic evaluation of the patient to identify possible risk factors for forming recurrent stones, which consists of a 24 hour urine analysis to determine the content of urinary components such as calcium or oxalate that play a major role in stone disease. High levels of oxalate and calcium contribute to kidney stones recurrences and therapy to reduce these two substances in the urine can reduce recurrence rates. Low levels of citrate also increase the risk for forming stones, and can be treated with alkali such as potassium citrate.

Collecting 24-hour urines for evaluation and therapy can be cumbersome for patients and often leads to incorrect collection, which may be detectable by measuring the amount of creatinine in each sample. Previous attempts to evaluate spot versus 24-hour urines have been made, but more studies are necessary to determine how they compare to the conventional 24-hour collection. A more convenient method for collecting urine samples will facilitate the treatment and future prevention of recurrent kidney stone disease.

The aim of this project is to determine whether spot urines collected separately at key times throughout the day are comparable to the conventional pooled 24-hour urine collection, and whether the former yield more accurate information in terms of the levels of urinary components. Perhaps a patient with normal values for a pooled 24-hour collection may show spikes in certain variables throughout the day that would not be discovered in the 24-hour sample. Furthermore, reducing the collection to a single time point would improve patient compliance making it easier to do subsequent follow-up collections.

HYPOTHESIS AND OBJECTIVES We hypothesize that spot urines can provide equivalent information to that provided by a 24-hour urine test. An added benefit would be if spot urines provide more information for the identification of risk factors in patients who have normal 24-hour urine tests. A third possibility is that our hypothesis is incorrect and that a 24-hour urine sample will provide the most useful data in formulating a stone prevention therapy for our patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed as having calcium based urinary stones
* at least 19 years of age
* do not have any additional serious disease

Exclusion Criteria:

* Patients who do not have calcium based urinary stones (such as: uric acid, cystine, struvite)
* less than 19 years of age
* have a serious alternate disease
* Pregnancy
* Positive Urine Culture
* Active cancer
* Recurrent urinary infections
* Gross hematuria
* Receiving treatment with thiazides (or alternatively can be enrolled if the patient is willing to stop treatment for 2 weeks prior to study)
* Inability to provide informed consent
* Investigator's refusal to include

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving care at Vancouver General Hospital for their kidney stone disease.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2009-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Calcium supersaturation and the risk of Calcium Oxalate crystallization will be compared between individual spot urines and conventional 24-hour urine sample | 24 hours divided into 4 time frames (spot urines)

SECONDARY OUTCOMES:
Identified risk factors for kidney stone patients will be compared between individual spot urines and conventional 24-hour urine sample: volume, pH, Urinary calcium, magnesium, oxalate, citrate, creatinine | 24 hours divided in 4 time frames (spot urines)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Paterson, Study Director — University of British Columbia; Roger Sutton, Study Director — University of British Columbia; Morris Pudek, Study Director — University of British Columbia; Dirk Lange, Study Director — University of British Columbia; Meredith Cushing, Study Director — Vancouver General Hospital
Locations (1):
- Vancouver General Hospital, DHCC, Level 6, 2775 Laurel Street, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No